CLINICAL TRIAL: NCT05680883
Title: Better Control and Treatment of Ulcerative Colitis by Exploring the Universe of Microenvironment Imposed Tissue Signatures and Their Correlates in Liquid Biopsies
Brief Title: Local and Systemic Immunoprofiling of Patients Diagnosed With Ulcerative Colitis
Acronym: ImmUniverse
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL78552.091.21
Record Dates: First submitted 2022-11-17; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-11

CONDITIONS: Ulcerative Colitis Flare
Keywords: Immune cells; Inflamed + non-inflamed biopsies + correlated blood samples; Flow cytometry; IHC; Single cell RNA sequencing; Immunoprofiling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — EDTA Whole Blood (3x 10mL) and colonic biopsies (4 inflamed and 4 uninflamed)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Immune-mediated diseases are extremely diverse - patients with the same diagnosis may see the disease progress in very different ways, and respond differently to treatments. This is because the course of the disease is influenced by multiple factors, including the patient's genes, immune system, environment, and the microbes living in their gut. Furthermore, all of these factors interact with and impact on one another. As a result, it is very hard to predict how the disease will develop in a specific patient, and which treatments will be effective. Hence, mechanistic understanding of this heterogeneity and biomarkers predictive for disease control and therapy response over time are important prerequisites of a future precision medicine in IMIDs. ImmUniverse has been formed as a European transdisciplinary consortium to tackle these unmet needs and to understand the role of the crosstalk between tissue microenvironment and immune cells in disease progression and response to therapy of ulcerative colitis (UC) and atopic dermatitis (AD).

The consortium will combine analysis of tissue-derived signatures with "circulating signatures" detectable in liquid biopsies, employing state-of-the-art profiling technologies to provide new validated diagnostics in IMID that are expected to improve patient management, lead to increased patient well-being and will significantly reduce the socioeconomic burden of these diseases. This study, being Immuniverse work package 5 (WP5), will verify the disease pathway -and mechanism signatures identified in the multi omic discovery WP2 in immune cells in affected tissue and peripheral blood. WP5 aims to further substantiate our understanding of the immune-mediated intestinal disease ulcerative colitis (UC). It will use liquid biopsies (peripheral blood) and affected UC gut inflamed and non-inflamed biopsies to generate transcriptome, proteome, DNA-methylome and miRNA signatures of immune cell subsets and analyse the association between immune cells circulating in peripheral blood and the microenvironment of affected colonic tissue.

Also this WP aims to develop a protocol to analyse and sort living immune cells from cryopreserved tissue. Ultimately, the project's findings should contribute to a better, more precise diagnosis for patients; and better information on how severe the disease is likely to be for each individual patient and how it will progress over time. Finally, the project will make it easier for doctors and patients to monitor how well a treatment is working in the future.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ulcerative Colitis
* Age ≥ 18 years
* Present in the hospital for a regular outpatient visit
* Willing and able to comply with the study related procedures
* Provide signed informed consent

Exclusion Criteria:

* Age ≤ 18 years
* Unable to give informed consent
* Unable or unwilling to comply with study-related procedures
* Crohn's Disease or IBD undiagnosed

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: 40 adult participants diagnosed with Ulcerative colitis and treated at the department of gasteroenterology of the Radboudumc.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-11-05 (Estimated); Study Completion 2023-11-05 (Estimated)

PRIMARY OUTCOMES:
Comparing immune cells in blood, inflamed and uninflamed colonic biopsies by means of flow cytometry | Through study completion, an average of 1.5 years
  Assessed by differences in Mean Fluorescent Intensity in whole blood sampels vs. inflamed and uninflamed biopsies
Comparing immune cells in blood, inflamed and uninflamed colonic biopsies by means of flow cytometry | Through study completion, an average of 1.5 years
  Assessed by differences in percentages of cell populations in whole blood sampels vs. inflamed and uninflamed biopsies
Comparing gene expression profiles in blood, inflamed and uninflamed colonic biopsies | Through study completion, an average of 1.5 years
  Assessment of mean expression of genes in blood vs. inflamed and uninflamed biopsies by means of single cell RNA sequencing
Localizing immune cells of interest of inflamed and uninflamed biopsies | Through study completion, an average of 1.5 years
  By using immunohistochemistry: quantified by cells per field

SECONDARY OUTCOMES:
For 40 patients: height | Through study completion, an average of 1.5 years
  Height in centimeter, combined with weight to get to BMI (kg/m^2)
For 40 patients: weight | Through study completion, an average of 1.5 years
  Weight in kilograms, combined with height to get to BMI (kg/m^2)
For 40 patients: smoking status | Through study completion, an average of 1.5 years
  1. Current/active smoker
  2. Previous smoker
  3. Never smoked
  4. Not described
For 40 patients: montreal classification | Through study completion, an average of 1.5 years
  1. E1: ulcerative proctitis
  2. E2: left-sided UC (distal to splenic flexure)
  3. E3: Entensive UC (pancolitis)
For 40 patients: SCCAI-score | Through study completion, an average of 1.5 years
  Based on 6 variables:
  1. Bowel frequency (day)
  2. Bowel frequency (night)
  3. Urgency of defecation
  4. Blood in stool
  5. General well-being
  6. Extracolonic features
For 40 patients: Mayo score (based on physician rating of endoscopic disease activity) | Through study completion, an average of 1.5 years
  0: normal or inactive disease
  1: mild disease (erythema, decreased vascular pattern, mild friability) 2. Moderate disease (marked erythema, absent vascular pattern, friability, erosions) 3. Severe disease (spontaneous bleeding, ulcerations)
For 40 patients: Medication history and current medication | Through study completion, an average of 1.5 years
  anti-TNF, Vedolizumab, Janus kinase inhibitors, thiopurine, methotrexate, aminosalicylates, corticosteroids (grams of medication/day)
For 40 patients: Feacel calprotectin | Through study completion, an average of 1.5 years
  mg/kg feces
For 40 patients: Albumin | Through study completion, an average of 1.5 years
  g/L
For 40 patients: infections in stool | Through study completion, an average of 1.5 years
  yes/no
Blood parameters | Through study completion, an average of 1.5 years
  WBC count (*10^9/L), RBC count (*10^12/L), PLT (*10^9/L), Lymphocytes (*10^9/L), Monocytes (*10^9/L), Neutrophils (*10^9/L), Eosinophils (*10^9/L), Basiphils (*10^9/L)

CONTACTS AND LOCATIONS:
Locations (1):
- RadboudUMC, Nijmegen, Gelderland, Netherlands